CLINICAL TRIAL: NCT02091024
Title: Blood Lipid-lowering Effect of Brown Alga Ecklonia Cava Extract in Hypercholesterolemic Korean Subjects: a Randomized Double-blind, Placebo-controlled Clinical Trial
Brief Title: Blood Lipid-lowering Effect of Brown Alga Ecklonia Cava
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Chonbuk National University Hospital (Other)
Responsible Party: Principal Investigator, Soo-Wan Chae, Clinical Trial Center for Functional Food, Chonbuk National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: LVCM-HL-SEAPOLYNOL
Record Dates: First submitted 2014-03-17; First posted 2014-03-19 (Estimated); Last update posted 2014-03-19 (Estimated); Status verified 2014-03

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — Endothelin-Converting Enzymes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ECG (Ecklonia cava extract) (Experimental): ECE 200mg, twice a day
  Interventions: Dietary Supplement: ECE (Ecklonia cava extract)
- Placebo (Placebo Comparator): Placebo 200mg, twice a day
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: ECE (Ecklonia cava extract) — ECE 200mg, twice a day
  Arms: ECG (Ecklonia cava extract)
Dietary Supplement: Placebo — Placebo 200mg, twice a day
  Arms: Placebo

SUMMARY:
The investigators performed a 12-week, randomized, double-blind, placebo-controlled human trial to evaluate the efficacy and safety of Ecklonia cava extract on hyperlipidemia.

DETAILED DESCRIPTION:
The investigators performed a 12-week, randomized, double-blind, placebo-controlled human trial to evaluate the efficacy and safety of Ecklonia cava extract on hyperlipidemia. The investigators measured improvement of lipid profile, including total cholesterol, triglyceride, HDL-cholesterol, and LDL-cholesterol.

ELIGIBILITY:
Inclusion Criteria:

* Mild hypercholesterolemic subjects(≥200mg/dL of total cholesterol or ≥110mg/dL of LDL-cholesterol)

Exclusion Criteria:

* Self-reported pregnancy, lactation
* Prevalent heart disease, cancer, renal disorder, or diabetes mellitus, and use of lipid-lowering drugs

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2011-04; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Changes in total cholesterol | 12 weeks
Changes in LDL-cholesterol | 12 weeks

SECONDARY OUTCOMES:
Changes in triglyceride | 12 weeks
Changes in HDL-cholesterol | 12 weeks
Changes in waist to hip ratio | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trial Center for Functional Foods; Chonbuk National University Hospital, Jeonju, Jeollabuk-do, South Korea